CLINICAL TRIAL: NCT01734200
Title: Efficacy and Safety of Eriobotyra Japonica Lindley Extract on Improvement of Cognitive Function: a 12 Week, Randomized Double-blind, Placebo-controlled Clinical Trial
Brief Title: Efficacy and Safety of Eriobotyra Japonica Lindley Extract on Improvement of Cognitive Function
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Chonbuk National University Hospital (Other)
Responsible Party: Principal Investigator, Soo-Wan Chae, Principal Investigator, Clinical Trial Center for Functional Foods, Chonbuk National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: INs-MF-ERIO
Record Dates: First submitted 2012-11-22; First posted 2012-11-27 (Estimated); Last update posted 2015-07-15 (Estimated); Status verified 2015-07

CONDITIONS: Cognitive Function

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Eriobotyra Japonica Lindley Extract (Experimental)
  Interventions: Dietary Supplement: Eriobotyra Japonica Lindley Extract
- Placebo (Placebo Comparator)
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Eriobotyra Japonica Lindley Extract — Eriobotyra Japonica Lindley Extract (1.5g/day)
  Arms: Eriobotyra Japonica Lindley Extract
Dietary Supplement: Placebo — Placebo (1.5g/day)
  Arms: Placebo

SUMMARY:
The investigators performed a 12-week, randomized, double-blind, placebo-controlled human trial to evaluate the efficacy and safety of Eriobotyra Japonica Lindley Extract on improvement of Memory Function. The investigators measured decrement of improvement of Memory Function, including K-MMSE, Rey-Kim Memory Test, BCRS, and PRMQ, and monitored their blood pressure.

ELIGIBILITY:
Inclusion Criteria:

* Males and females 16-19 years old
* Weight within ±30% of ideal body weight
* Able to give informed consent

Exclusion Criteria:

* Allergic or hypersensitive to any of the ingredients in the test products
* History of reaction to any of the test products or of gastrointestinal diseases such as Crohn's disease or gastrointestinal surgery
* History of alcohol or substance abuse
* Participation in any other clinical trials within past 2 months
* Laboratory test, medical or psychological conditions deemed by the investigators to interfere with successful participation in the study
* Pregnant or lactating women etc.

Ages: 16 Years to 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 80 (Actual)
Dates: Start 2012-11; Primary Completion 2013-09 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Changes in K-MMSE(Korean Mini-Mental State Examination) | 12 weeks
  K-MMSE(Korean Mini-Mental State Examination) was measured in study visit 1(0 week) and visit 3(12 week).

SECONDARY OUTCOMES:
Changes in Rey-Kim Memory Test | 12 weeks
  Rey-Kim Memory Test was measured in study visit 1(0 week) and visit 3(12 week).
Changes in BCRS(Brief Cognitive Rating Scale) | 12 weeks
  BCRS(Brief Cognitive Rating Scale) was measured in study visit 1(0 week) and visit 3(12 week).
Changes in PRMQ(Prospective and retrospective memory questionnaire) | 12 weeks
  PRMQ(Prospective and retrospective memory questionnaire) was measured in study visit 1(0 week) and visit 3(12 week).
Changes in STAI(State-trait anxiety inventory) | 12 weeks
  STAI(State-trait anxiety inventory) was measured in study visit 1(0 week) and visit 3(12 week).
Changes in BDNF(Brain derived neurotrophic factor) | 12 weeks
  BDNF(Brain derived neurotrophic factor) was measured in study visit 1(0 week) and visit 3(12 week).

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical Trial Center for Functional Foods; Chonbuk National University Hospital, Jeonju, Jeollabuk-do, South Korea